CLINICAL TRIAL: NCT00620295
Title: Phase I Study of Bortezomib and Gemcitabine in Elderly Patients With Solid Tumors (X05227)
Brief Title: Bortezomib and Gemcitabine in Treating Older Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000586510; UMN-2006LS040 (Other: CPRC, University of Minnesota); UMN-X05227 (Other: Millennium Pharm., Inc.); x464 (Other: Eli Lilly & Co.)
Record Dates: First submitted 2008-02-20; First posted 2008-02-21 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Head and Neck Cancer; Kidney Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Sarcoma
Keywords: recurrent pancreatic cancer; recurrent breast cancer; recurrent small cell lung cancer; recurrent non-small cell lung cancer; recurrent colon cancer; recurrent prostate cancer; recurrent head and neck cancer; ovarian cancer; recurrent uterine cancer; recurrent kidney cancer; recurrent osteosarcoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Sarcoma; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Uterine Neoplasms; Osteosarcoma | interventions — Bortezomib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine / Bortezomib (Experimental): Gemcitabine will be administered as a 30 minute intravenous infusion at the patient's assigned dose on day 1 and day 8 of a 21 day cycle.
  Bortezomib will be given 1 hour after gemcitabine by IVP over 3 to 5 seconds followed by a standard saline on days 1 and 8 of a 21 day treatment cycle until disease progression or for a maximum of 6 cycles.
  Interventions: Drug: bortezomib; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: bortezomib — Bortezomib will be given 1 hour after gemcitabine by intravenous pyelogram (IVP) over 3 to 5 seconds followed by a standard saline flush or through a running intravenous (IV) line at the patient's assigned dose (1.0 up to 1.8 mg/m^2) on days 1 and 8 of a 21 day treatment cycle until disease progression or for a maximum of 6 cycles.
  Other Names: Velcade
Drug: gemcitabine hydrochloride — Gemcitabine will be administered as a 30 minute intravenous infusion at the patient's assigned dose (800 up to 1000 mg/m^2) on day 1 and day 8 of a 21 day cycle.
  Other Names: Gemzar

SUMMARY:
RATIONALE: Bortezomib may stop the growth of solid tumors by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with gemcitabine may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib and gemcitabine in treating older patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of weekly bortezomib and gemcitabine in treating elderly patients with advanced solid tumors.

Secondary

* To characterize the quantitative and qualitative toxicities of bortezomib and gemcitabine in these patients.
* To obtain preliminary information about the anti-tumor activity of bortezomib and gemcitabine.
* To characterize gemcitabine and metabolite pharmacokinetics in patients receiving concurrent bortezomib therapy.

OUTLINE: This is a phase I dose escalation study of bortezomib and gemcitabine.

Patients receive gemcitabine intravenously (IV) over 30 minutes followed 1 hour later by bortezomib IV over 3-5 seconds on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine and bortezomib until the maximum tolerated dose of the combination is determined.

Blood is collected periodically for pharmacokinetic and pharmacogenetic studies.

After completion of study treatment, patients are followed every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced non-hematologic malignancy, including any of the following:

  * Breast cancer
  * Lung cancer
  * Colon cancer
  * Pancreatic cancer
  * Head and neck cancer
  * Sarcoma
* Must have failed or become intolerant to prior standard therapy and is no longer likely to respond to such therapy (for all diseases except pancreatic cancer)

  * Pancreatic cancer patients may be enrolled with no prior therapy requirements since gemcitabine is the current standard of care 1st line therapy
* Measurable or nonmeasurable disease
* Concurrent enrollment in the University of Minnesota study "Population Pharmacokinetics and Pharmacogenetics of Gemcitabine in Adult Patients with Solid Tumors" (Human Subjects Code 0508M72989) required
* ECOG performance status of 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3.0 times ULN (5 times ULN if liver has tumor involvement)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 times ULN (5 times ULN if liver has tumor involvement)
* Calculated or measured creatinine clearance > 30 mL/minute
* Fertile patients must use effective contraception during and for 3 months after study participation
* Recovered from all prior therapy
* Prior systemic chemotherapy, immunotherapy, or biological therapy allowed
* At least 3 months since prior bortezomib and/or gemcitabine
* At least 2 weeks since prior systemic therapy
* At least 3 weeks since prior investigational agents (for reasons other than the treatment of cancer)
* At least 2 weeks since prior radiotherapy

Exclusion Criteria:

* Symptomatic brain metastases
* Serious concomitant medical or psychiatric disorders (e.g., active infection or uncontrolled diabetes) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* Myocardial infarction within the past 6 months
* New York Heart Association (NYHA) Class III or IV heart failure
* Uncontrolled angina
* Severe uncontrolled ventricular arrhythmias
* Electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Peripheral neuropathy ≥ grade 2
* Known hypersensitivity to bortezomib, boron or mannitol
* Prior radiotherapy to ≥ 25% of the bone marrow
* Prior radiotherapy to the whole pelvis
* Concurrent filgrastim (G-CSF) or other hematologic support during course 1 of study treatment

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib and gemcitabine | Day 21 (Week 3 - Cycle 1)
  A minimum of a 3 week period (1 cycle) must be completed by all patients within a dose level before dose escalation to the next level may occur. A cycle is defined as treatment day 1 and 8 with follow-up through day 21.

SECONDARY OUTCOMES:
Toxicity | 30 Days after Last Treatment
  Toxicity will be graded using the NCI's Common Terminology Criteria for Adverse Events (CTCAE 3.0)
Disease response as measured by RECIST criteria | Week 4
  The best overall response is the best response recorded from the start of treatment until disease progression/recurrence, taking as reference for progressive disease the smallest measurements recorded since the treatment began.
Characterization of gemcitabine and metabolite pharmacokinetics (as part of co-enrollment in Population Pharmacokinetics and Pharmacogenetics of Gemcitabine in Adult Patients with Solid Tumors") | Pre-Dose
  Pharmacokinetics will be done in conjunction with the dosing day 1 of cycle 1 whenever possible.

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States